CLINICAL TRIAL: NCT00314678
Title: Cisplatin Induction Followed by Paclitaxel Consolidation for the Treatment of Stage III and IV Epithelial Ovarian Cancer and Primary Peritoneal Cancer With In Vitro Correlates of Response
Brief Title: Cisplatin Induction With Paclitaxel Consolidation for Stage III-IV Epithelial Ovarian and Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: John P. Fruehauf (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, John P. Fruehauf, Dr. John P. Fruehauf, University of California, Irvine
Organization: University of California, Irvine (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 99-25
Record Dates: First submitted 2006-04-12; First posted 2006-04-14 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2007-12

CONDITIONS: Epithelial Ovarian Cancer; Primary Peritoneal Cancer
Keywords: Ovarian; Peritoneal
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Topotecan; Cisplatin; Paclitaxel

INTERVENTIONS:
Drug: Topotecan
Drug: Cisplatin
Drug: Paclitaxel

SUMMARY:
Clinically, there has been extensive experience with topotecan and cisplatin. Recently, several investigators have evaluated the combination of paclitaxel, cisplatin and topotecan. As expected, myelosuppression was the dose-limiting factor. Herben et al recently reported the results of a phase I trial using the combination of paclitaxel, cisplatin, and topotecan as first line therapy in advanced stage ovarian cancer. Interestingly, the authors could not achieve a dose of topotecan that would be considered "optimal" for the treatment of relapsed disease in a single-agent fashion. The inability to utilize a therapeutic dose when combined with either platinum or paclitaxel has been demonstrated in previous reports and affirms the bone marrow suppressive effect. The clinical response rate from this trial was reported as 86.7%.

DETAILED DESCRIPTION:
Malignant neoplasms of the ovary are the cause of more deaths than any other gynecologic cancer. Approximately 26,500 new cases are diagnosed each year in the United States, and about 14,500 deaths occur annually as a result of this disease. Clinicians continue to be frustrated by both the paucity of data concerning the etiologic factors in epithelial ovarian cancer and by the failure to achieve a significant reduction in mortality over the past several decades.

Since the introduction of cisplatin-based chemotherapy, no treatment has been shown to improve survival in subjects with advanced ovarian cancer until the incorporation of paclitaxel into primary therapy for this disease. In 1996, the Gynecologic Oncology Group (GOG) published the results of a large prospective, randomized trial of cisplatin and cyclophosphamide compared to cisplatin and paclitaxel. The cisplatin plus paclitaxel regimen was noted to be superior based on: 1) an overall improved response rate; 2) an increased clinical response rate (51% vs. 31%); 3) an increased rate of negative second look laparotomies; 4) an increase in median progression free survival; and importantly 5) an increased overall median survival (38 months vs. 24 months). The GOG results were recently confirmed by the Canadian- European consortium randomized phase III trial (OV 10).

These large randomized trials established the combination of paclitaxel and cisplatin as the standard, first line therapy for women with advanced ovarian cancer following cytoreductive surgery. Although the majority of women with advanced ovarian cancer will demonstrate an objective response to this combination; the response is generally of limited duration. The five-year survival for advanced stage ovarian cancer is 20-40%. Consequently, there remains a need for an improved chemotherapeutic approach in the management of ovarian cancer.

Topotecan is a semi-synthetic analog of camptothecin, a topoisomerase inhibitor. It has been investigated in a number of phase II trials as salvage therapy for recurrent ovarian cancer. Overall response rates have ranged from 6% to 27%. In a randomized comparative trial of topotecan versus paclitaxel, overall response rates were 21% and 14% respectively. The median survival for topotecan was 63 weeks as compared to 53 weeks for paclitaxel. Both drugs demonstrated higher response rates in platinum-sensitive tumors than platinum-resistant tumors. These data suggest that topotecan may be as active as paclitaxel, and partially non-cross resistant with cisplatin.

Topotecan may be a better agent than paclitaxel for use in combination with cisplatin for multiple reasons. First, Kern et al demonstrated that paclitaxel may antagonize the activity of cisplatin. Second, topotecan has been demonstrated to be synergistic with both cisplatin and paclitaxel in vitro. It has been demonstrated that topotecan can dramatically potentiate the effects of platinum, perhaps by its ability to inhibit repair of platinum-DNA adducts.

Clinically, there has been extensive experience with topotecan and cisplatin. Recently, several investigators have evaluated the combination of paclitaxel, cisplatin and topotecan. As expected, myelosuppression was the dose-limiting factor. Herben et al recently reported the results of a phase I trial using the combination of paclitaxel, cisplatin, and topotecan as first line therapy in advanced stage ovarian cancer. Interestingly, the authors could not achieve a dose of topotecan that would be considered "optimal" for the treatment of relapsed disease in a single-agent fashion. The inability to utilize a therapeutic dose when combined with either platinum or paclitaxel has been demonstrated in previous reports and affirms the bone marrow suppressive effect. The clinical response rate from this trial was reported as 86.7%.

ELIGIBILITY:
Eligible Subjects:

1. Subjects with a histologic diagnosis of epithelial ovarian cancer or primary peritoneal carcinoma, stage III or IV, as outlined above. All subjects must have appropriate surgery for ovarian carcinoma with appropriate tissue for histologic evaluation and evaluated by the EDR assay.
2. Eligible cell types include:

   Serous adenocarcinoma Endometrioid adenocarcinoma Mucinous adenocarcinoma Undifferentiated carcinoma Clear cell adenocarcinoma Mixed epithelial carcinoma Transitional cell carcinoma Malignant Brenner's Tumor
3. Adequate bone marrow, renal, and hepatic function as defined by WBC3000cells/mcl, platelets 100,000/mcl, serum creatinine 2mg/dcl, bilirubin 1.5times normal, and SGOT 3 times normal.
4. Subjects with GOG Performance Status of 0, 1, or 2.
5. Subjects must have a complete history and physical examination done by the investigators of this study. Also, CBC with differential, electrolytes, serum creatinine, liver function tests and CA 125 must be done 14 days prior to registration.
6. Subjects must be informed of the investigational nature of this study and must provide informed consent in accordance with institutional and federal guidelines.
7. All subjects must have histologic slides available for pathology review.
8. Subjects must be entered within six weeks of surgery.

Ineligible Subjects:

1. Subjects with epithelial ovarian carcinoma of low malignant potential.
2. Subjects who have received prior radiotherapy or chemotherapy.
3. Subjects with septicemia, severe infection, or acute hepatitis.
4. Subjects with severe gastrointestinal bleeding.
5. Subjects with a GOG Performance Status of 3 or 4.
6. Subjects with other invasive malignancies, with the exception of non-melanoma skin cancer, who had or have any evidence of other cancer within the last 5 years or whose previous cancer treatment contradicts this protocol therapy.
7. Subjects who are pregnant will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2005-09; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Recurrence-Free Interval

SECONDARY OUTCOMES:
Examine the toxicity of therapy and to develop suitable strategies for dose modification.

CONTACTS AND LOCATIONS:
Overall Officials: John P Fruehauf, MD, PhD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States